CLINICAL TRIAL: NCT04216394
Title: Anticoagulation in Emergency General Surgery: Who Bleeds More? The ACES Trial
Brief Title: Anticoagulation in Emergency General Surgery
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 049.GME.2019.D
Record Dates: First submitted 2019-11-27; First posted 2020-01-02 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-02

CONDITIONS: Emergency General Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Emergency general surgery — multidisciplinary surgery performed for traumatic and non-traumatic acute conditions during the same admission in the hospital.

SUMMARY:
While DOACs are increasing in use in the EGS patient population, the risk of bleeding and the reversal of these agents to reduce hemorrhage is still evolving. Given the paucity of data regarding the impact of DOACs in this patient population, it becomes empiric to identify bleeding patterns and outcomes in the EGS population taking DOACs. We hypothesize that patients taking a DOAC will have a higher bleeding incidence and need for an unplanned intervention secondary to hemorrhage in EGS patients undergoing an urgent or emergent operation when compared to patients taking warfarin and antiplatelets.

DETAILED DESCRIPTION:
Emergency general surgery (EGS) represents illnesses of diverse pathology with urgent/emergent treatment needs being the common denominator.A characteristic feature of EGS is its limitation in patient preparation. It is difficult and often impossible to eliminate certain patient dependent factors to reduce the operative risk. It has been reported that the annual case rate in the EGS population is (1,290 per 100,000) higher than the sum of all cancer diagnoses. The EGS burden is substantial and continues to increase. The elderly patient population represents 48% of the overall EGS population. With the increase in the prevalence of atherosclerotic disease in the elderly there has been an increase in the use of antiplatelets and anticoagulants.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are confirmed to be taking dabigatran, rivaroxaban, apixaban, warfarin and antiplatelet therapy (aspirin, clopidogril, ticagrelor) undergoing an urgent or emergent surgical intervention by the emergency general surgery service within 24 hours of arrival to the hospital
* 18 years of age or over

Exclusion Criteria:

* Prisoners
* Pregnant patients
* Those who received an index operation at an outside facility and were transferred
* Under 18 years of age

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Emergency general surgery patient population taking Direct oral anticoagulants
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2020-11-13 (Actual)

PRIMARY OUTCOMES:
Rate of operative | Oct 2019 - Aug 2021
  To determine the bleeding risk and need for unplanned intervention
Number of Participants with interventional radiology | Oct 2019 - Aug 2021
  To determine the bleeding risk and need for unplanned intervention
Number of Participants with ultrasound aspiration | Oct 2019 - Aug 2021
  To determine the bleeding risk and need for unplanned intervention

CONTACTS AND LOCATIONS:
Overall Officials: Michael Truitt, MD, Principal Investigator — Methodist Dallas Medical Center Trauma
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided